CLINICAL TRIAL: NCT00442572
Title: Stop Progression of Fibrosis by Administration of Intermittent Continuous Treatment With Peginterferon Alfa-2a. Open-label, Randomized Efficacy and Safety Clinical Trial of Intermittent Continuous Treatment With Peginterferon Alfa-2a (PEGASYS) in Patients With HBeAg Negative Hepatitis B Responding to Prior Treatment With Interferon Alfa (SOFIA -LTT)
Brief Title: SOFIA-LTT Study: A Study of Intermittent Long Term Treatment With PEGASYS (Peginterferon Alfa-2a (40KD)) in Patients With HBeAg Negative Chronic Hepatitis B (CHB).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML20020
Record Dates: First submitted 2007-02-15; First posted 2007-03-02 (Estimated); Results first posted 2016-04-11 (Estimated); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a

ARMS (2):
- PEGASYS (Experimental): Participants received 4 treatment cycles of continuous intermittent treatment with PEGASYS® (Peginterferon alfa-2a) . Each cycle consisted of 12 weeks injection treatment with Peginterferon alfa-2a 135 micrograms in 0.5 ml solution in prefilled syringes, applied once weekly subcutaneously and followed by 12 weeks period without treatment.
  Interventions: Drug: PEGASYS [peginterferon alfa-2a]
- No Intervention (No Intervention): Participants were on non- specific anti-viral treatment.

INTERVENTIONS:
Drug: PEGASYS [peginterferon alfa-2a] — There were 4 treatment cycles of continuous intermittent treatment with Peginterferon alfa-2a. Each cycle consisted of 12 weeks injection treatment with Peginterferon alfa-2a 135 micrograms in 0.5 ml solution in prefilled syringes, applied once weekly subcutaneously and followed by 12 weeks period without treatment.
  Arms: PEGASYS

SUMMARY:
This 2 arm study will evaluate the efficacy and safety of intermittent treatment with PEGASYS in HBeAg negative patients with chronic hepatitis B who have demonstrated virological and biochemical response after treatment with interferon alfa. After 48 weeks therapy with interferon alfa, and 24 weeks treatment-free follow-up, eligible patients will be randomized into the PEGASYS or the observational group. Those in the PEGASYS group will receive 4 therapeutic cycles of long term intermittent treatment with PEGASYS (135 micrograms sc weekly for 12 weeks, followed by a treatment-free period of 12 weeks) and those in the observational arm will receive no specific antiviral treatment. The anticipated time on study treatment is 1-2 years, and the target sample size is 100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* liver disease consistent with CHB;
* evidence of chronic HBeAg-negative CHB prior to initial course of interferon alfa;
* patients who have responded to previous 48 weeks treatment with interferon alfa.

Exclusion Criteria:

* coinfection with HCV, HDV or HIV;
* decompensated liver disease, hepatocellular cancer, or evidence of a medical condition associated with chronic liver disease other than viral hepatitis;
* any other systemic antiviral, antineoplastic or immunomodulatory treatment <=6 months prior to first dose of randomized treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2006-07-03 (Actual); Primary Completion 2012-04-23 (Actual); Study Completion 2012-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Mhat St. Ivan Rilski; Clinic of Gastroenterology, Sofia, Bulgaria

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants in this study were enrolled at one centre in Bulgaria from 03 July 2006 to 23 April 2012. Of the 21 participants enrolled, 17 participants were randomized to PEGASYS arm and 4 participants were randomized to no intervention arm.
Groups:
- PEGASYS: Participants received 4 treatment cycles of continuous intermittent treatment with Peginterferon alfa-2a (PEGASYS®). Each cycle consisted of 12 weeks injection treatment with Peginterferon alfa-2a 135 micrograms (µg) in 0.5 ml solution in prefilled syringes, applied once weekly subcutaneously (SC) and followed by 12 weeks period without treatment.
Period: Overall Study
Arm/Group | PEGASYS | No Intervention
Started | 17 | 4
Completed | 9 | 1
Not Completed | 8 | 3
Not completed — Relapse | 8 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all the randomized participants who passed during at least one treatment period, and had at least one efficacy and safety evaluation.
Groups:
- PEGASYS: Participants received 4 treatment cycles of continuous intermittent treatment with Peginterferon alfa-2a. Each cycle consisted of 12 weeks injection treatment with Peginterferon alfa-2a 135 µg in 0.5 ml solution in prefilled syringes, applied once weekly SC and followed by 12 weeks period without treatment.
- Total: Total of all reporting groups
Arm/Group | PEGASYS | No Intervention | Total
Number analyzed (Participants) | 17 | 4 | 21
Age, Continuous [Median (Full Range); unit: years] | 44 [23 to 61] | 38.5 [22 to 50] | 42 [22 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 0 | 7
  Male | 10 | 4 | 14

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Stable Virological Response
Description: Stable virological response is serum Hepatitis B virus deoxyribonucleic acid (HBV DNA) <20 000 copies/ml during the treatment (after each 12 weeks) and after the follow-up period (24 weeks after the last treatment period).
Time Frame: Up to Week 108
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | PEGASYS | No Intervention
Number analyzed (Participants) | 17 | 3
Percentage of Participants
  Week 12 | 100 [80.49 to 100.00] | 100.0 [29.24 to 100.00]
  Week 24 | 52.9 [27.81 to 77.02] | 66.7 [9.42 to 99.16]
  Week 36 | 52.9 [27.81 to 77.02] | 100.0 [29.24 to 100.00]
  Week 48 | 47.1 [22.98 to 72.19] | 66.7 [9.42 to 99.16]
  Week 60 | 47.1 [22.98 to 72.19] | 33.3 [0.84 to 90.58]
  Week 72 | 41.2 [18.44 to 67.08] | 33.3 [0.84 to 90.58]
  Week 84 | 41.2 [18.44 to 67.08] | 33.3 [0.84 to 90.58]
  Week 96 | 29.4 [10.31 to 55.96] | 33.3 [0.84 to 90.58]
  Week 108 | 29.4 [10.31 to 55.96] | 33.3 [0.84 to 90.58]

2. Secondary Outcome: Percentage of Participants With Stable Virological and Biochemical Response
Description: All participants who achieved virological response (serum HBV DNA < 20 000 copies/ml) and biochemical response (stable normalization of their alanine transaminase [ALT]) during the treatment cycle (after each 12 weeks) and after the follow-up period (24 weeks after the last treatment period).
Time Frame: Up to Week 108
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | PEGASYS | No Intervention
Number analyzed (Participants) | 17 | 3
Percentage of Participants
  Week 12 | 100.0 [80.49 to 100.00] | 100.0 [29.24 to 100.00]
  Week 24 | 52.9 [27.81 to 77.02] | 66.7 [9.42 to 99.16]
  Week 36 | 52.9 [27.81 to 77.02] | 100.0 [29.24 to 100.00]
  Week 48 | 47.1 [22.98 to 72.19] | 66.7 [9.42 to 99.16]
  Week 60 | 47.1 [22.98 to 72.19] | 33.3 [0.84 to 90.58]
  Week 72 | 41.2 [18.44 to 67.08] | 33.3 [0.84 to 90.58]
  Week 84 | 41.2 [18.44 to 67.08] | 33.3 [0.84 to 90.58]
  Week 96 | 29.4 [10.31 to 55.96] | 33.3 [0.84 to 90.58]
  Week 108 | 29.4 [10.31 to 55.96] | 33.3 [0.84 to 90.58]

3. Secondary Outcome: Percentage of Participants With Loss of Hepatitis B Surface Antigen
Description: Loss of Hepatitis B Surface Antigen (HBsAg) was defined as change of detectable HBsAg from positive to negative.
Time Frame: Up to Week 108
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | PEGASYS | No Intervention
Number analyzed (Participants) | 17 | 3
Percentage of Participants | 5.9 [0.14 to 28.69] | 0 [0 to 0]

4. Secondary Outcome: Percentage of Participants With HBsAg Seroconversion
Description: The development of antibodies against HBsAg is known as HBsAg seroconversion. It signifies clearance of HBsAg and resolution of the chronic infection. НBsAg seroconversion is the final goal of anti-hepatitis B virus treatment and it is closest to the definition of "cure" but in practice it is very rare in HBeAg-negative chronic hepatitis B (CHB).
Time Frame: Up to Week 108
Population: Safety population included all the randomized participants who passed during at least one treatment period, and had at least one efficacy and safety evaluation. Data of participants available at the time of the assessment were included in the analysis. Only participants with HBsAg clearance were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | PEGASYS | No Intervention
Number analyzed (Participants) | 1 | 0
Percentage of Participants | 0 |

5. Secondary Outcome: Percentage of Participants With HBV DNA Levels Under the Lower Limit (Serum HBV DNA Level < 300 Copies/ml) For a Significant Quantity
Description: HBV DNA level, or viral load, is an indicator of viral replication. Higher HBV DNA levels are usually associated with an increased risk of liver disease and hepatocellular carcinoma. HBV DNA level typically falls in response to effective antiviral treatment.
Time Frame: Up to Week 108
Population: Safety population included all randomized participants who passed during at least one treatment period and had at least one efficacy and safety evaluation. HBV DNA levels below lower limit for significant quantity were not studied for no intervention arm participants.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | PEGASYS | No Intervention
Number analyzed (Participants) | 17 | 0
Percentage of Participants | 29.4 [10.3 to 56.0] |

6. Secondary Outcome: Fibrosis-4 and Aspartate Aminotransferase to Platelet Ratio Index Scores For Change in Liver Fibrosis
Description: Fibrosis-4 (FIB-4) and Aspartate Aminotransferase to Platelet Ratio Index (APRI) are non-invasive scoring systems, which are calculated on the basis of laboratory tests that indicates the level of liver fibrosis. The APRI scores are calculated based on Aspartate Aminotransferase (AST) levels and platelet counts whereas FIB-4 scores are calculated based on platelets, ALT, AST and age. For APRI, the scores are interpreted as ≤ 0.5 is 81% sensitive and 50% specific for a diagnosis of significant fibrosis in chronic hepatitis C (CHC), where as a cut-off > 1.5 is 35% sensitive and 91% specific for the diagnosis of significant fibrosis. The majority of biomarker panels will produce inconclusive results for a proportion of participants falling within the indeterminate range (between 0.5 and 1.5) for a specific fibrosis end-point. For FIB-4, the scores are interpreted as FIB-4 score of < 1.45: absence of cirrhosis, FIB-4 score of 1.45 to 3.25: inconclusive, FIB-4 score > 3.25: cirrhosis.
Time Frame: Up to Week 108
Population: as for baseline characteristics
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | PEGASYS | No Intervention
Number analyzed (Participants) | 13 | 0
Units on a scale
  FIB-4 | 1.06 [0.36 to 2.66] |
  APRI | 0.25 [0.14 to 1.48] |

7. Secondary Outcome: Mean Change From Baseline in HBsAg Levels
Description: An early decrease in HBsAg from baseline to Weeks 12 or 24 has been identified as further on-treatment predictor for sustained HBsAg clearance and virological response in HBeAg negative participants.
Time Frame: Up to Week 108
Population: Safety population included all the randomized participants who passed during at least one treatment period, and had at least one efficacy and safety evaluation. Data of participants available at the time of the assessment were included in the analysis.
Measure: Mean (95% Confidence Interval); unit: copies/mL
Arm/Group | PEGASYS | No Intervention
Number analyzed (Participants) | 17 | 3
copies/mL
  Week 12, n=17,3 | -1156.00 [-5212.33 to 2900.33] | -240.50 [-3715.65 to 3234.65]
  Week 24, n=17,3 | -1293.72 [-5756.89 to 3169.45] | -146.00 [-7172.53 to 6880.53]
  Week 36, n=14,3: number analyzed (Participants) | 14 | 3
  Week 36, n=14,3 | -3049.64 [-7949.30 to 1850.01] | -564.00 [-4248.80 to 3120.80]
  Week 48, n=13, 3: number analyzed (Participants) | 13 | 3
  Week 48, n=13, 3 | -1591.78 [-9217.83 to 6034.28] | -528.50 [-2987.15 to 1930.15]
  Week 60, n=11,1: number analyzed (Participants) | 11 | 1
  Week 60, n=11,1 | -3096.56 [-11135.37 to 4942.26] | -379.00 [NA to NA] — For Week 60, only one participant had valid data based on which 95% CI cannot be constructed.
  Week 72, n=10, 1: number analyzed (Participants) | 10 | 1
  Week 72, n=10, 1 | -3485.90 [-10299.06 to 3327.26] | -34.00 [NA to NA] — For Week 72, only one participant had valid data based on which 95% CI cannot be constructed.
  Week 84, n=9, 1: number analyzed (Participants) | 9 | 1
  Week 84, n=9, 1 | 201.40 [-11899.81 to 12302.61] | -54.72 [NA to NA] — For Week 84, only one participant had valid data based on which 95% CI cannot be constructed.
  Week 96, n=14,1: number analyzed (Participants) | 14 | 1
  Week 96, n=14,1 | -3011.75 [-8046.71 to 2023.21] | -49.51 [NA to NA] — For Week 96, only one participant had valid data based on which 95% CI cannot be constructed.
  Week 108, n=12,0: number analyzed (Participants) | 12 | 0
  Week 108, n=12,0 | -3368.13 [-7625.12 to 888.87] |

8. Secondary Outcome: Mean Change From Baseline in Hemoglobin
Description: The hemoglobin values were planned to be calculated as arithmetic mean by treatment groups (PEGASYS and No Intervention).
Time Frame: Up to Week 108
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Gram/deciliter
Arm/Group | PEGASYS | No Intervention
Number analyzed (Participants) | 12 | 0
Gram/deciliter | -1.73 (10.44) |

9. Secondary Outcome: Mean Change From Baseline in Hematology
Description: The hematology parameters included erythrocytes, leucocytes, basophils, eosinophils, lymphocytes, monocytes, thrombocytes. All laboratory parameters were planned to be calculated as arithmetic mean by treatment groups (PEGASYS and No Intervention).
Time Frame: Up to Week 108
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | PEGASYS | No Intervention
Number analyzed (Participants) | 12 | 0
10^9/L
  Erythrocytes | 0.08 (0.26) |
  Leukocytes | -1.72 (2.00) |
  Basophils | -0.18 (0.38) |
  Lymphocytes | 5.56 (6.31) |
  Monocytes | 1.87 (3.10) |
  Thrombocytes | -31.20 (36.40) |
  Eosinophils | 0.92 (1.24) |

10. Secondary Outcome: Mean Change From Baseline in Clinical Chemistry
Description: The clinical chemistry parameters included alanine aminotransferase (ALAT), aspartate aminotransferase (ASAT), gamma-glutamyl transferase (GGT), alkaline phosphatase (ALP). All laboratory parameters were planned to be calculated as arithmetic mean by treatment groups (PEGASYS and No Intervention).
Time Frame: Up to Week 108
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Units/Litre
Arm/Group | PEGASYS | No Intervention
Number analyzed (Participants) | 12 | 0
Units/Litre
  ALAT | 5.56 (25.44) |
  ASAT | 9.00 (27.76) |
  GGT | 1.00 (3.70) |
  ALP | 50.92 (38.00) |

11. Secondary Outcome: Mean Change From Baseline in Protein and Indirect Albumin
Description: The clinical chemistry parameters included indirect protein and albumin. All laboratory parameters were planned to be calculated as arithmetic mean by treatment groups (PEGASYS and no intervention).
Time Frame: Up to Week 108
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Gram/deciliter
Arm/Group | PEGASYS | No Intervention
Number analyzed (Participants) | 12 | 0
Gram/deciliter
  Protein indirect | -31.62 (38.70) |
  Albumin | -1.35 (1.71) |

12. Secondary Outcome: Mean Change From Baseline in Bilirubin Indirect and Bilirubin Direct
Description: The laboratory parameters included bilirubin indirect and bilirubin direct. All laboratory parameters were planned to be calculated as arithmetic mean by treatment groups (PEGASYS and No Intervention).
Time Frame: Up to Week 108
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: milligrams/deciliter
Arm/Group | PEGASYS | No Intervention
Number analyzed (Participants) | 12 | 0
milligrams/deciliter
  Indirect bilirubin | -0.95 (3.38) |
  Direct bilirubin | -0.16 (0.77) |

13. Secondary Outcome: Mean Change From Baseline in Blood Urea
Description: The blood urea was planned to be calculated as arithmetic mean by treatment groups (PEGASYS and No Intervention).
Time Frame: Up to Week 108
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: millimoles/liter
Arm/Group | PEGASYS | No Intervention
Number analyzed (Participants) | 12 | 0
millimoles/liter | -0.34 (1.23) |

14. Secondary Outcome: Mean Change From Baseline in Creatinine and Uric Acid
Description: The creatinine and uric acid values were planned to be calculated as arithmetic mean by treatment groups (PEGASYS and No Intervention).
Time Frame: Up to Week 108
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: micromole/liter
Arm/Group | PEGASYS | No Intervention
Number analyzed (Participants) | 12 | 0
micromole/liter
  Creatinine | -3.65 (13.23) |
  Uric acid | -21.51 (130.42) |

15. Secondary Outcome: Mean Change From Baseline in Blood Glucose
Description: The blood glucose was measured for change from baseline. All blood glucose values were planned to be calculated as arithmetic mean by treatment groups (PEGASYS and No Intervention).
Time Frame: Up to Week 108
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: millimoles/ liter
Arm/Group | PEGASYS | No Intervention
Number analyzed (Participants) | 12 | 0
millimoles/ liter | -0.06 (0.40) |

16. Secondary Outcome: Mean Change From Baseline in Thyroid Stimulating Hormone (TSH)
Description: The TSH was planned to be calculated as arithmetic mean by treatment groups (PEGASYS and No Intervention).
Time Frame: Up to Week 108
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: milli-international units/liter
Arm/Group | PEGASYS | No Intervention
Number analyzed (Participants) | 12 | 0
milli-international units/liter | 0.67 (1.50) |

17. Secondary Outcome: Mean Change From Baseline in Triiodothyronine and Thyroxine
Description: The Triiodothyronine (T3) and thyroxine (T4) values were planned to be calculated as arithmetic mean by treatment groups (PEGASYS and No Intervention).
Time Frame: Up to Week 108
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: picomole/liter
Arm/Group | PEGASYS | No Intervention
Number analyzed (Participants) | 12 | 0
picomole/liter
  T3, Week 108 | 0.19 (5.44) |
  T4, Week 108 | -0.85 (4.99) |

ADVERSE EVENTS:
Time Frame: Up to Week 108
Description: AE is untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is with any of the following outcomes: Death, initial or prolonged inpatient hospitalization, life-threatening experience, persistent or significant disability/incapacity; congenital anomaly.
Groups:
- PEGASYS: Participants received 4 treatment cycles of continuous intermittent treatment with Peginterferon alfa-2a. Each cycle consisted of 12 weeks injection treatment with Peginterferon alfa-2a 135 micrograms in 0.5 ml solution in prefilled syringes, applied once weekly subcutaneously and followed by 12 weeks period without treatment.
Arm/Group | PEGASYS | No Intervention
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/4
Other Adverse Events (participants affected / at risk) | 11/17 | 1/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PEGASYS (N=17) | No Intervention (N=4)
Muscle pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Joint ache (Musculoskeletal and connective tissue disorders) | 1 | 0
Adjustment disorder with mixed anxiety and depressed mood (Psychiatric disorders) | 1 | 0
Allergic Rhinitis (Immune system disorders) | 1 | 0
Tonsilllitis bacterial (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Dental and gingival conditions (Gastrointestinal disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 0
Dysmenorrhea (Reproductive system and breast disorders) | 2 | 0
Expectoration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Fatigue (General disorders) | 2 | 0
Hair loss (Skin and subcutaneous tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 1
Herpes simplex (Infections and infestations) | 2 | 0
Hypertonia (Vascular disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Nausea and vomiting symptoms (Gastrointestinal disorders) | 1 | 0
Open wound of knee, leg (except thigh), and ankle, without mention of complication (Surgical and medical procedures) | 1 | 0
Pyrexia (General disorders) | 3 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Stomach ache (Gastrointestinal disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.